CLINICAL TRIAL: NCT06244719
Title: Vibrotactile Stimulation for Neurological Disorders
Brief Title: Vibrotactile Stimulation for Upper-Extremity Stroke Rehabilitation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-0783
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibrotactile Stimulation (Experimental): Participants wear vibrotactile stimulation shirts and gloves for 5 hours per day, 7 days per week, during their stay at the rehabilitation unit, which is expected to be between 2-3 weeks. Participants wear the devices after conventional therapy is done for the day.
  Interventions: Device: Vibrotactile Stimulation
- Control (No Intervention): Participants undergo conventional therapy only.

INTERVENTIONS:
Device: Vibrotactile Stimulation — Shirts contain embedded vibration motors that stimulate the impaired upper-extremity at 18 different locations. The gloves stimulates the fingertips.
  Arms: Vibrotactile Stimulation

SUMMARY:
The goal of this clinical trial is to investigate upper-extremity vibrotactile stimulation with wearables in stroke patients. The main questions it aims to answer are:

Are the wearables well-tolerated by patients? Does the vibrotactile stimulation help regain arm function?

Participants will wear vibrotactile stimulation gloves and shirts for 5 hours daily during their stay at the rehabilitation unit, in addition to conventional therapy. Researchers will compare the treatment group (vibrotactile stimulation wearables) with a control group (conventional therapy only) to see the effects of the vibrotactile stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at rehabilitation units
* Unilateral left or right sided ischemic stroke within the previous 2 weeks
* Have Upper-Extremity Fugl-Meyer scores between 6 and 58
* Have at least 20 degrees of active shoulder elevation and elbow flexion
* Expected to stay 1-3 weeks in the rehabilitation unit

Exclusion Criteria:

* Under anti-spasticity therapy
* Patients that are dependent on pacemakers
* Patients that have defibrillators
* Have lymphedema or AV fistula for dialysis on an arm

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Test of Sensorimotor Function After Stroke (UEFM) | Baseline, End of the study (approximately 1-3 weeks, at discharge from the rehabilitation unit).
  An impairment based measure consisting of 33 movements that tests motor and sensation of the affected arm. Higher scores indicate less impairment and more isolated motions. Scores are between 0 and 66.

SECONDARY OUTCOMES:
Number of participants with at least one adverse event | End of the study (approximately 1-3 weeks, at discharge from the rehabilitation unit).
  Adverse event will only include those that are determined to be related to the vibrotactile stimulation
Number of participants who completed the therapy | End of the study (approximately 1-3 weeks, at discharge from the rehabilitation unit).
  Vibrotactile stimulation therapy feasibility will be assessed by the number of participants who completed the therapy
Number of participants who tolerated the vibrotactile stimulation therapy | End of the study (approximately 1-3 weeks, at discharge from the rehabilitation unit).
  Therapy tolerability will be assessed by responses to questionnaires
Change in the modified Ashworth scale | Baseline, End of the study (approximately 1-3 weeks, at discharge from the rehabilitation unit).
  The modified Ashworth scale is used to assess spasticity and tests the resistance to passive movement about a joint with varying degree of velocity. The modified Ashworth scale assigns a grade of spasticity from a 0-4 ordinal scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCHealth Rehabilitation Unit, Aurora, Colorado
  - Broomfield Hospital, Broomfield, Colorado

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06244719/Prot_SAP_000.pdf